CLINICAL TRIAL: NCT00664963
Title: YUKON-drug-eluting Stent Below The Knee - Prospective Randomized Double-blind Multicenter Study
Brief Title: YUKON-drug-eluting Stent Below The Knee - Randomised Double-blind Study
Acronym: YUKON-BTK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Thomas Zeller, Prof., Herz-Zentrums Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YUKON-BTK v3.0
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Arterial Occlusive Diseases
Keywords: Arterial Occlusive Diseases; Peripheral Vascular Diseases; Drug eluting stent; Restenosis; Below the knee; Intervention
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): YUKON Sirolimus-eluting Stent
  Interventions: Device: Implantation of YUKON Sirolimus-eluting Stent
- 2 (Active Comparator): YUKON Stent (uncoated)
  Interventions: Device: Implantation of YUKON Stent (uncoated)

INTERVENTIONS:
Device: Implantation of YUKON Sirolimus-eluting Stent — Implantation of YUKON Sirolimus-eluting Stent
  Arms: 1
Device: Implantation of YUKON Stent (uncoated) — Implantation of YUKON Stent (uncoated)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of the treatment with balloon-expandable YUKON-BTX-Sirolimus-eluting stent over the treatment with YUKON-BTX uncoated stent in patients with ischemic infrapopliteal arterial disease.

DETAILED DESCRIPTION:
Based on the fact that drug eluting stents have been proven to reduce the restenosis rate in the coronary arteries, we assume that YUKON-BTX-Sirolimus-eluting stent has a superior restenosis rate compared to treatment with uncoated stent in the below-the-knee arteries consecutively. The purpose of this study is to compare the restenosis rate of the treatment with balloon-expandable YUKON-BTX-Sirolimus-eluting stent over the treatment with YUKON-BTX uncoated stent in patients with ischemic infrapopliteal arterial disease. Randomisation will be performed by extremity, that may lead to varying treatments within one patient during the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of peripheral arterial occlusive disease as defined by Rutherford 2-5
* De-novo stenosis of > 70% diameter stenosis in the tibioperoneal trunc, anterior and/or posterior tibial and/or peroneal artery
* Target lesion length of ≤ 45 mm

Exclusion Criteria:

* Coagulation disorder
* Known allergy to contrast medium
* Contraindications to antiplatelet therapy or heparin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Restenosis rate after 12 months (> 50% stenosis by angiography or duplex ultrasound) | 12 months

SECONDARY OUTCOMES:
Number of reinterventions of target vessel | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Herz-Zentrum Bad Krozingen
Locations (3):
- Germany (3):
  - Herz-Zentrums Bad Krozingen, Bad Krozingen
  - Universitäres Herzzentrum Hamburg, Hamburg
  - University Hospital of Tübingen, Tübingen

REFERENCES:
- [Derived] Rastan A, Brechtel K, Krankenberg H, Zahorsky R, Tepe G, Noory E, Schwarzwalder U, Macharzina R, Schwarz T, Burgelin K, Sixt S, Tubler T, Neumann FJ, Zeller T. Sirolimus-eluting stents for treatment of infrapopliteal arteries reduce clinical event rate compared to bare-metal stents: long-term results from a randomized trial. J Am Coll Cardiol. 2012 Aug 14;60(7):587-91. doi: 10.1016/j.jacc.2012.04.035. PMID 22878166
- [Derived] Rastan A, Tepe G, Krankenberg H, Zahorsky R, Beschorner U, Noory E, Sixt S, Schwarz T, Brechtel K, Bohme C, Neumann FJ, Zeller T. Sirolimus-eluting stents vs. bare-metal stents for treatment of focal lesions in infrapopliteal arteries: a double-blind, multi-centre, randomized clinical trial. Eur Heart J. 2011 Sep;32(18):2274-81. doi: 10.1093/eurheartj/ehr144. Epub 2011 May 26. PMID 21622669